CLINICAL TRIAL: NCT02445274
Title: Effectiveness of Two Different Surgical Procedures to Prevent Posterior Capsule Opacification in Age-related Cataract Patients
Brief Title: Two Different Cataract Surgical Procedures to Prevent Posterior Capsule Opacification
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Associate Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015MEKY046
Record Dates: First submitted 2015-05-04; First posted 2015-05-15 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Cataract; Posterior Capsule Opacification
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capsule-reserved surgical procedure (Experimental): In this group, the anterior lens capsule was reserved after continuous curvilinear capsulorhexis. The reserved anterior capsule was pressed flattened by the optical surface of the IOL and attached onto the posterior lens capsule.
  Phacoemulsification was performed with the same device and handpieces, using the same phaco chop technique as in the conventional procedure group.
  Interventions: Procedure: Anterior lens capsule was reserved
- Conventional surgical procedure (No Intervention): In this group, the anterior lens capsule was not reserved or attached onto the posterior lens capsule.

INTERVENTIONS:
Procedure: Anterior lens capsule was reserved — The anterior lens capsule was reserved after continuous curvilinear capsulorhexis. The reserved anterior capsule was pressed flattened by the optical surface of the IOL and attached onto the posterior lens capsule.
  Arms: Capsule-reserved surgical procedure

SUMMARY:
In this study, the investigators introduce a new "capsule-reserved" cataract surgical procedure in which anterior lens capsule is reserved and attached onto posterior lens capsule in the purpose of preventing posterior capsule opacification (PCO). A prospective randomized controlled study is reported to compare the new "capsule-reserved" surgical procedure with conventional one on the effectiveness to prevent posterior capsule opacification in age-related cataract patients.

DETAILED DESCRIPTION:
A prospective, randomized controlled study of 240 eligible patients will been enrolled. Two eyes of each patient were assigned randomly to two groups respectively: Group I; anterior lens capsule is conventionally not reserved after continuous curvilinear capsulorhexis, while in Group II, anterior lens capsule is innovatively reserved and attached onto posterior lens capsule. This novel adjusted surgical procedure, featured by using the reserved anterior lens capsule to protect the peri-capsule microenvironment and prevent PCO, is conceptual different from the traditional cataract surgical procedure. Clinical examinations including posterior capsule opacification grading score, central posterior capsule thickness, central posterior capsule density, best corrected visual acuity, contrast sensitivity were carried out preoperatively and at each postoperative visit.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 50 years or above
2. Both eyes were diagnosed with age-related cataract
3. Both eyes were planed to undergo the "Phacoemulsification and IOL implantation" surgery with 1 month
4. Biocular BCVA improvement post surgery was feasible judged by the ophthalmologists.

Exclusion Criteria:

1. Other ocular diseases
2. ACD<3CT
3. Combined cataract surgery (trabeculoplasty, keratoplasty)
4. Lens pseudoexfoliation syndrome combined with glaucoma or zonular abnormalities
5. Previous intraocular surgery or trauma (laser not included)
6. Uveitis
7. Recent ocular infection
8. Proliferative diabetic retinopathy
9. Diabetes mellitus
10. Congenital ocular abnormalities (aniridia, congenital cataract)
11. Atrophy of iris
12. Participants with previous clinical trials 30 days before surgery
13. Using prostanoid eye drops
14. Uncontrolled systematic diseases

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in posterior capsule opacification grading score | post-operative day 1, post-operative week 1, post-operative month 1, post-operative month 3,
  Posterior capsule opacification（PCO）was recorded by standardized slit lamp retroillumination images and analyzed using the EPCO2000 program. The severity of PCO was clinically graded from 0 (none) to 4 (severe)

SECONDARY OUTCOMES:
Change from Baseline in central posterior capsule thickness | post-operative day 1, post-operative week 1, post-operative month 1, post-operative month 3, post-operative month 6, post-operative year 1
  Central posterior capsule thickness was recorded and calculated by Pentacam HR system
Change from Baseline in central posterior capsule density | post-operative day 1, post-operative week 1, post-operative month 1, post-operative month 3, post-operative month 6, post-operative year 1
  Central posterior capsule density was recorded and calculated by Pentacam HR system.

OTHER OUTCOMES:
Change from Baseline in best corrected visual acuity | post-operative day 1, post-operative week 1, post-operative month 1, post-operative month 3, post-operative month 6, post-operative year 1
  Best-corrected visual acuity (BCVA) was measured, using an ETDRS chart and auto-refraction as refined by an ophthalmologist.
Change from Baseline in contrast sensitivity | post-operative day 1, post-operative week 1, post-operative month 1, post-operative month 3, post-operative month 6, post-operative year 1
  Contrast sensitivity under mesopic and photopic conditions was measured using C-quant

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, M.D., PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Luo L, Lin H, Chen W, Qu B, Zhang X, Lin Z, Chen J, Liu Y. Intraocular lens-shell technique: adjustment of the surgical procedure leads to greater safety when treating dense nuclear cataracts. PLoS One. 2014 Nov 17;9(11):e112663. doi: 10.1371/journal.pone.0112663. eCollection 2014. PMID 25401512
- [Background] Lin H, Yan P, Yu K, Luo L, Chen J, Lin Z, Chen W. Anterior segment variations after posterior chamber phakic intraocular lens implantation in myopic eyes. J Cataract Refract Surg. 2013 May;39(5):730-8. doi: 10.1016/j.jcrs.2012.12.026. Epub 2013 Mar 14. PMID 23499067
- [Background] Lin HT, Chen WR, Ding ZF, Chen W, Wu CR. Clinical evaluation of two multifocal intraocular lens implantation patterns. Int J Ophthalmol. 2012;5(1):76-83. doi: 10.3980/j.issn.2222-3959.2012.01.16. Epub 2012 Feb 18. PMID 22553760
- [Result] Luo L, Lin H, He M, Congdon N, Yang Y, Liu Y. Clinical evaluation of three incision size-dependent phacoemulsification systems. Am J Ophthalmol. 2012 May;153(5):831-839.e2. doi: 10.1016/j.ajo.2011.10.034. Epub 2012 Feb 4. PMID 22310081
- See also: Homepage for Zhongshan Ophthalmic Center — http://www.gzzoc.com